CLINICAL TRIAL: NCT03631290
Title: Deprescribing for Older Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00100184; 1K76AG059930 (NIH)
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-11

CONDITIONS: Kidney Failure, Chronic
Keywords: kidney failure, chronic; renal dialysis; aged; inappropriate prescribing; preliminary data
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who were approached to undergo deprescribing: If the patient's nephrologist agreed to attempt deprescribing the PIM, either the nephrologist (Provider Only Communication) or a study team member (pharmacist or nurse, Provider/Patient Communication) would engage the patient in discussion about deprescribing.
  Interventions: Behavioral: Deprescribing Intervention
- Providers: Nephrologists and Advanced Practice Providers who see patients at a Duke affiliated DaVita hemodialysis (HD) clinic where Duke nephrologists serve as medical directors and rounding physicians

INTERVENTIONS:
Behavioral: Deprescribing Intervention — The deprescribing program was implemented as a clinical quality improvement project for patients receiving dialysis. Patients taking specific potentially inappropriate medications (PIMs) were identified in the medical record. The PIMs of interest included gabapentinoids, clonidine, alpha blockers, muscle relaxants, and Z-drugs. If their nephrologist agreed to attempt deprescribing the PIM, either the nephrologist (Provider Only Communication) or a study team member (pharmacist or nurse, Provider/Patient Communication) would engage the patient in discussion about deprescribing. This discussion included patient education materials about the risk of the medication. If the patient agreed, they were provided taper instructions (if indicated) and were followed up at 1 month and 3 months.
  The patient was also invited to enroll in a study to be interviewed about the deprescribing decision and experience, and undergo brief assessment of geriatric problems at baseline and at 3 months.
  Groups: Patients who were approached to undergo deprescribing

SUMMARY:
Aim 1 of the study is to identify the elements of a deprescribing intervention that address contextual factors specific to dialysis.

Aim 2 of the study, described in this record, is to determine the feasibility of a deprescribing intervention tailored for older dialysis patients.

Older adults receiving dialysis are often prescribed multiple medications. Some of these medications are used to treat symptoms, but they also can increase the chance of significant health problems. The purpose of this study is to identify if it is feasible to reduce the use of medications that have been identified as causing an increased risk for health problems.

ELIGIBILITY:
Inclusion Criteria (patients):

* an adult receiving dialysis for at least 6 months
* at least one active prescription for a potentially inappropriate medication (gabapentinoids, clonidine, alpha blockers, muscle relaxants, and Z-drugs)

Exclusion Criteria (patients):

* advanced dementia
* hospice care
* non-English speaking

Inclusion Criteria (providers):

* must be employed by Duke
* must see patients at a Duke affiliated DaVita hemodialysis (HD) clinic where Duke nephrologists serve as medical directors and rounding physicians

Exclusion Criteria (providers):

None

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient participants include community-dwelling hemodialysis patients. Providers will be Nephrologists and Advanced Practice Providers who are members of the Deprescribing QIP team at Duke-affiliated DaVita Dialysis clinics.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rasheeda K Hall, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not assigned to an arm upon entry. The study assessed two distinct approaches to shared decision-making: Provider Communication Only and Provider/Patient Communication. The purpose of the study was to assess feasibility of deprescribing overall and not to compare the two approaches. Therefore, participant data is only reported by decision-making group where practicality of Provider/Patient Communication was assessed.
  Providers were assessed as one group.
Period: Overall Study
Arm/Group | Patients Who Were Approached to Undergo Deprescribing | Providers
Started | 41 | 7
Participants Who Agreed to Deprescribe | 17 | 0
Completed | 41 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Who Were Approached to Undergo Deprescribing | Providers | Total
Number analyzed (Participants) | 41 | 7 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was not collected from Providers
  years
    number analyzed (Participants) | 41 | 0 | 41
    (all) | 67.2 (8.1) |  | 67.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 2 | 21
  Male | 22 | 5 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 40 | 0 | 40
  Unknown or Not Reported | 0 | 7 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 32 | 0 | 32
  White | 8 | 0 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 7 | 7
Region of Enrollment [Number; unit: participants]
  United States | 41 | 7 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Deprescribing Events
Description: Deprescribing events will be assessed for the Provider Only and Provider/Patient communication approaches. While this data is categorized into the two approaches, it is not intended for comparison.
Time Frame: 3 months
Population: 34 participants were Provider Only, and 7 were Provider/Patient Communication.
Measure: Number; unit: deprescribing events
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 41
deprescribing events
  Provider Only Communication: number analyzed (Participants) | 34
  Provider Only Communication | 15
  Provider/Patient Communication: number analyzed (Participants) | 7
  Provider/Patient Communication | 2

2. Primary Outcome: Number of Potentially Eligible Subjects
Description: The study team identified patients aged 55 and older with active prescriptions for specific potentially inappropriate medications (PIMs) (gabapentinoids, clonidine, alpha blockers, muscle relaxants, and Z-drugs) from the medical record and met criteria for deprescribing.
Time Frame: Baseline
Population: Total number of potentially eligible participants are reported. Not all potentially eligible participants were enrolled in the study.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Potentially Eligible Participants: The study team identified patients aged 55 and older with active prescriptions for specific potentially inappropriate medications (PIMs) (gabapentinoids, clonidine, alpha blockers, muscle relaxants, and Z-drugs) from the medical record and met criteria for deprescribing.
Arm/Group | Number of Potentially Eligible Participants
Number analyzed (Participants) | 85
Participants | 85

3. Primary Outcome: Proportion of Clinicians Who Found the Deprescribing Program Met Their Approval
Description: This is an assessment of provider acceptability, defined as those who answered "agree" or "completely agree" to the Likert item: The deprescribing program meets my approval.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Providers
Number analyzed (Participants) | 7
Participants | 5

4. Primary Outcome: Proportion of Clinicians Who Found the Deprescribing Program Fit Their Routine
Description: This is an assessment of provider acceptability. The outcome was defined as those who answered "agree" or "completely agree" to the Likert item: The deprescribing program seems fitting with my clinical routine.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Providers
Number analyzed (Participants) | 7
Participants | 2

5. Primary Outcome: Proportion of Clinicians Who Found the Deprescribing Program Seemed Doable
Description: This is an assessment of provider acceptability. The outcome was defined as those who answered "agree" or "completely agree" to the Likert item: The deprescribing program seems doable.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Providers
Number analyzed (Participants) | 7
Participants | 5

6. Secondary Outcome: Number of Adverse Drug Withdrawal Events
Description: Symptoms develop related to cutting back or stopping a medication. This was identified by chart review and/or if reported by patient to study team.
Time Frame: 3 months
Population: Only participants who agreed to deprescribe were assessed for adverse drug withdrawal events.
Measure: Number; unit: events
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 17
events | 7

7. Secondary Outcome: Change in Functional Assessment
Description: Enrolled participants completed the Older Americans Resources and Services (OARS) functional assessment which assesses instrumental and basic activities of daily living (ADLs). The instrument scores range from 0-28, with higher scores indicating better ability to do ADLs.
Time Frame: Baseline, 3 months
Population: Of those approached, this subset agreed to complete assessments at the time of decision and 3 months after decision for deprescribing. This subset includes all individuals irrespective of their deprescribing decision (yes or no).
Measure: Mean (Standard Error); unit: change in score on OARS assessment
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 11
change in score on OARS assessment | 1.27 (0.47)

8. Secondary Outcome: Change in Fall Risk Questionnaire
Description: Enrolled participants completed the CDC STEADI Fall Risk instrument. The instrument scores range from 0-14, with higher scores indicating a greater risk of falls.
Time Frame: Baseline, 3 months
Population: as for outcome 7
Measure: Mean (Standard Error); unit: change in score in CDC STEADI Fall Risk
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 11
change in score in CDC STEADI Fall Risk | -0.3 (0.4)

9. Secondary Outcome: Change in Patient Health Questionnaire-9 (PHQ9)
Description: Enrolled participants completed the PHQ9 instrument which assesses for depression. The instrument scores range from 0-27, with higher scores indicating a greater depression severity.
Time Frame: Baseline, 3 months
Population: as for outcome 7
Measure: Median (Standard Error); unit: change in score on PHQ9
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 11
change in score on PHQ9 | -1.36 (1.08)

10. Secondary Outcome: Change in Cognitive Change Index
Description: Enrolled participants completed the Cognitive Change Index instrument which assesses for cognition. The instrument scores range from 0-100, with higher scores indicating a greater likelihood of cognitive impairment.
Time Frame: Baseline, 3 months
Population: as for outcome 7
Measure: Mean (Standard Error); unit: change in cognitive change index score
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 11
change in cognitive change index score | -2.8 (10.8)

11. Secondary Outcome: Sustainability, as Measured by the Proportion of Patients Who Remained Off PIM at a Lower Dose
Description: Among those who deprescribed, the study team followed up by phone to inquire if they were still off the PIM and/or taking a lower dose than before
Time Frame: 3 months
Population: only 6 participants were available for 3 month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 6
Participants | 4

12. Secondary Outcome: Practicality, as Measured by Average Time (in Days) Spent Awaiting Provider Response to Deprescribing Recommendation
Description: The investigators will compare practicality of Provider-only Communication and Provider/Patient Communication because the Provider/Patient Communication involved additional staff outside of the dialysis clinic and such staff would not be guaranteed in real-world application of this intervention.
Time Frame: Baseline
Population: 34 participants were Provider Only, and 7 were Provider/Patient Communication.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 41
days
  Provider-only: number analyzed (Participants) | 34
  Provider-only | 10 [5 to 32]
  Provider/Patient Communication: number analyzed (Participants) | 7
  Provider/Patient Communication | 15 [5 to 43]

13. Secondary Outcome: Practicality, as Measured by the Average Time (in Days) to Initial Patient Communication
Description: The investigators will assess practicality in the QIP - Provider / Patient Communication format.
Time Frame: Baseline
Population: Analysis is limited to the 7 participants in the Provider/Patient Communication group.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 7
days | 21 [7 to 30]

14. Secondary Outcome: Practicality, as Measured by the Average Number of Attempts to Reach the Patient
Description: The investigators will assess practicality in the QIP - Provider / Patient Communication format.
Time Frame: Baseline
Population: Analysis is limited to the 7 participants in the Provider/Patient Communication group
Measure: Mean (Standard Deviation); unit: number of attempts
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 7
number of attempts | 4.3 (2.3)

15. Secondary Outcome: Practicality, as Measured by the Average Number of Conversations
Description: The investigators will assess practicality in the QIP - Provider / Patient Communication format.
Time Frame: Baseline
Population: Analysis is limited to the 7 participants in the Provider/Patient Communication group
Measure: Mean (Standard Deviation); unit: number of conversations
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 7
number of conversations | 1.4 (0.8)

16. Secondary Outcome: Practicality, as Measured by the Average Length of Conversations With Patients About Deprescribing
Description: The investigators will assess practicality in the QIP - Provider / Patient Communication format.
Time Frame: Baseline
Population: Analysis is limited to the 7 participants in the Provider/Patient Communication group
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Patients Who Were Approached to Undergo Deprescribing
Number analyzed (Participants) | 7
minutes | 13.6 (6.9)

ADVERSE EVENTS:
Time Frame: Within 1 month of starting to deprescribe the medication.
Description: Adverse Drug Withdrawal Events (ADWEs) include a physiological withdrawal reaction or intolerance of deprescribing (worsened symptoms). ADWEs were collected for patients who were approached to undergo deprescribing, agreed to deprescribe, and then reported intolerance of cutting back or stopping the medication. No adverse events were collected from provider participants or patients who did not agree to undergo deprescribing.
Arm/Group | Patients Who Were Approached to Undergo Deprescribing | Providers
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/0
Other Adverse Events (participants affected / at risk) | 7/17 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients Who Were Approached to Undergo Deprescribing (N=17) | Providers (N=0)
Intolerance of deprescribing (Nervous system disorders) | 7 | 0 — Intolerance of deprescribing includes worsening or return of symptoms. Because the medications deprescribed addressed pain, we associate these ADWE with the Nervous Systems organ system.

LIMITATIONS AND CAVEATS:
This ClinicalTrials.gov record and results are specific to Aim 2 of the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03631290/Prot_SAP_000.pdf